CLINICAL TRIAL: NCT04646343
Title: Cross-cultural Adaptation and Validation of the "Cold Intolerance Symptom Severity Questionnaire" (CISS) and the "Potential Work Exposure Scale" (PWES) in Patients With Hand Pathologies.
Brief Title: Cross-cultural Adaptation and Validation of the CISS and the PWES Questionnaire in Patients With Hand Pathologies.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinique Romande de Readaptation (Network)
Responsible Party: Sponsor
Other Study IDs: CliniqueRR-08
Record Dates: First submitted 2020-11-11; First posted 2020-11-27 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2023-08

CONDITIONS: Hand Injuries and Disorders
Keywords: cold intolerance; questionnaire; cross cultural adaptation
MeSH Terms: conditions — Hand Injuries; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group for cross cultural adaptation of questionnaire: Pre final French version of the CISS and PWES will be administered to French native speaking patients suffering from various hand injuries. 30 patients are sufficient. They will be asked to write commentaries on difficulties of questionnaire's items, especially comprehension of the different items (clear or unclear).If the item is considered unclear, the patient is asked to provide suggestions for making the item clearer .The distribution of the responses will be examined for searching missing responses. An item considered unclear by 20 % or more of the patients must be re-evaluated . The definitive version of French-CISS and French PWES (F-CISS and F- PWES) and the verification of the different stages of the cross-cultural adaptation will be validated during a new consensus meeting.
  Interventions: Other: administration of F-CISS and F-PWES pre version
- group for validation of questionnaire: For the second part (validation study) we will administered F-CISS, F-PWES, F-DASH, F-HFS, F-SF 36 questionnaires and a pain VAS to a population of in and outpatients with hand injuries. We aim to include patients during one year for a total expected of 100 patients.
  Interventions: Other: administration of definitive version of F-CISS and F-PWES plus F-DASH, F-HFS and F-SF 36

INTERVENTIONS:
Other: administration of F-CISS and F-PWES pre version — the CISS questionnaire is a 6 items questionnaire, the PWES is a 3 items questionnaire. Only 10 minutes are required to fulfilled the questionnaires.
  Groups: group for cross cultural adaptation of questionnaire
Other: administration of definitive version of F-CISS and F-PWES plus F-DASH, F-HFS and F-SF 36 — The administration will required 25 minutes
  Groups: group for validation of questionnaire

SUMMARY:
The primary objective of the study is to do translation, cross-cultural adaptation and validation of the CISS and PWES questionnaire in French. No available translation exist in French.

In the first part of the study, the investigators will use clinical guidelines for translation and cross-cultural adaptation of questionnaire (Beaton and al).The content validity will be evaluated also in this first step.

In the second part of the study the French version of CISS and PWES (F-CISS and F-PWES) will be validated. Different psychometric properties (internal consistency, test retest reliability, construct validity, floor and ceiling effects) will be study. The investigators use the recommendation of COSMIN (COnsensus- based Standards for the selection of health Measurement INstruments) group.

DETAILED DESCRIPTION:
This study in the first part has a cross-cultural adaptation design. The investigators will use the CISS questionnaire modified by Ruijs, because the total score is between 0 and 100. For the PWES questionnaire the investigators will use the original version .For translation and cross-cultural adaptation, no consensus exists. The investigators choose the guidelines of AAOS outcomes committee which are widely used and accepted in the literature.

The following five steps will be documented in a written report: (1) forward translation from English to French by two translators whose native language is French and fluent in English (T1 and T2). One of the translators is informed about the aims of the study and the other received only limited information (so-called naive translator).Moreover, none of the translators are physicians. (2) Synthesis of T1 and T2 will be done to form a unique translated version T12 by resolving any discrepancies under supervision of a methodologist not involved in the translation process. (3) Back translation of the T12 version from French to English by two English native speaking who are fluent in French (BT1 and BT2). These two translators are naive to the study and not linked to the medical domain. (4) Consensus meeting with all the involved subjects (translators, methodologist, specialist physicians in rehabilitation) in order to resolve any discrepancies and doubts met during the translation and to establish the pre final French version of the CISS and PWES (5).

The investigators will verify content validity which is the ability to an instrument to reflect the domain of interest and the conceptual definition of a construct i.e. cold intolerance. For this purpose, the instructions, response format and the items of F-CIIS and F-PWES questionnaire will be evaluated by a panel of 10 people for conceptual equivalence (clarity). The expert panel will have knowledge's about the content areas of the construct of the questionnaire and the target population of the questionnaire. The mother language tongue of the expert panel is French. The experts have to rate if instructions, response format and items are clear or unclear. If unclear they are asked to provide suggestions for making the language clearer. If instructions, response format and items are found to be unclear by at least 20 % of the panel, they have to be revised. The minimum inter rater agreement among the experts panel is 80%.

Then the expert panel evaluate each item of the instrument for content equivalence, using the following scale (1=not relevant, 2=somewhat relevant, 3=quite relevant, 4=highly relevant). Items classified as 1 or 2 should be revised. Content validity index at the item level (I-CVI) and at the scale level (S-CVI) should be calculated. The averaging calculation of S-CVI (S-CVI/Ave) is the preferred method. With 10 experts, the I-CVI of 0.78 or above and an S-CVI/Ave of 0.90 or above are the minimum acceptable indices. Items that do not achieve the minimum acceptable indices are revised and re-evaluated.

This part of the study which not concerned patients run from November 2019 to September 2020.

Pre final French version of the CISS and PWES will be administered to French native speaking patients suffering from various hand injuries. 30 patients are sufficient[50]. They will be asked to write commentaries on difficulties of questionnaire's items, especially comprehension of the different items (clear or unclear).If the item is considered unclear, the patient is asked to provide suggestions for making the item clearer .An item considered unclear by 20 % or more of the patients must be re-evaluated . The definitive version of French-CISS and French PWES (F-CISS and F- PWES) and the verification of the different stages of the cross-cultural adaptation will be validated during a new consensus meeting.

For the second part (validation study) the investigators will administered F-CISS, F-PWES, F-DASH, F-HFS, F-SF 36 questionnaires and a pain VAS to a population of 100 in and outpatients with hand injuries. For F-CISS and F-PWES test-retest reliability, the first 50 patients consecutively included will be asked to answer questionnaires 7 days later .

The investigators propose to choose the cut-off of 30 points in the study to separate which patient has a CI or not.

For the second part of the study, validation, different statistics will be made.

For internal consistency:

Exploratory factor analysis: 7 to 10 subjects per item are recommended with preference for a sample ≥ 100 . To select the appropriate number of factors, many criteria might be used. We can look at the screeplot, or take all components with an eigenvalue > 1 (Kaiser Criterion). To interpret the factors, an orthogonal varimax rotation will be applied. After that, items will be associated with a given factor if their loadings are higher than 0.5 for the latter.

Calculation of Cronbach's α for the entire questionnaire and for the different dimensions. A Cronbach's α ≥0.70 for the entire questionnaire and for the subscales is required .

For test-retest reliability or reproducibility:

Intraclass Correlation Coefficient (ICC) are used. Since systematic difference is not expected between test and retest, a two-way random effect model will be applied, so that systematic difference are included in the measurement error. The investigators will study 50 patients with an interval of 7 days . The value of ICC should be >0.70 .

For construct validity: only the F-CISS will be studied. The F-PWES is only a scale for screening people which are exposed to cold in their work and doesn't explore the same dimensions. Pearson's correlation coefficient will be used.

Different hypotheses are posed.

1. The F-CIIS is well correlated with the F-DASH. A correlation ≥ 0.5 is expected.
2. The F-CISS is well correlated with the F-HFS. A correlation≥ 0.5 is expected.
3. The F-CISS is well correlated with pain VAS. A correlation ≥ 0.5 is expected. For pain VAS the question will be: when you are exposed to cold how much is your pain? We will use a 100 mm horizontal VAS.
4. The F-CISS is weakly correlated with SF36-PC. A correlation between 0.30 and 0.5 is expected.
5. The F-CISS is not associated with SF36-MC. A correlation < 0.3 is expected. To have a good construct validity, 75 % of the hypotheses should be satisfied .

Floor or ceiling effects: the distribution of scores will be observed and the investigators expected no floor or ceiling effects (less than 15 % of respondents achieved the highest or lowest possible scores).

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years.
* Hand injury or hand pathology with or without CRPS. The CRPS patients will have to meet the Budapest criteria
* Good French comprehension.

Exclusion Criteria

-Inability to follow the procedures of the study, e.g. due to language problems, severe psychological disorders, dementia, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the studied population will be in and out patients. Inpatients are patients hospitalized with hand injuries for a vocational rehabilitation in our clinic.. There are mainly men, with a mean age of 45 years, working in the secondary sector. All the patients which speak French will be invited to participate to the study.
  Outpatients are ambulatory patients seen in consultation with various hand problems (injuries or not). The mean age will be higher than in the first group and there will be more women. All the patients consulting for hand problems will be invited to participate to the study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of items of the two questionnaires considered as unclear by the patients | 3 months (February 2021)
  if more of 20 % of the patients considered item as unclear it should be revised
Percentage of patients with cold intolerance assessed by the CISS questionnaire | one year (December 2021)
  the cold intolerance is defined by a score more than 30 points (possible score from 0 to 100).

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Léger, PhD, Study Director — institut de recherche en réadaptatation
Locations (1):
- Clinique romande de réadaptation, Sion, Valais, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nancarrow JD, Rai SA, Sterne GD, Thomas AK. The natural history of cold intolerance of the hand. Injury. 1996 Nov;27(9):607-11. doi: 10.1016/s0020-1383(96)00110-6. PMID 9039355
- [Background] Vaksvik T, Hetland K, Rokkum M, Holm I. Cold hypersensitivity 6 to 10 years after replantation or revascularisation of fingers: consequences for work and leisure activities. J Hand Surg Eur Vol. 2009 Feb;34(1):12-7. doi: 10.1177/1753193408094440. Epub 2008 Dec 17. PMID 19091739
- [Background] Graham B, Schofield M. Self-reported symptoms of cold intolerance in workers with injuries of the hand. Hand (N Y). 2008 Sep;3(3):203-9. doi: 10.1007/s11552-008-9116-0. Epub 2008 Jul 3. PMID 18780096
- [Background] Carlsson IK, Nilsson JA, Dahlin LB. Cut-off value for self-reported abnormal cold sensitivity and predictors for abnormality and severity in hand injuries. J Hand Surg Eur Vol. 2010 Jun;35(5):409-16. doi: 10.1177/1753193409354184. Epub 2009 Dec 23. PMID 20031998
- [Background] Gustafsson M, Hagberg L, Holmefur M. Ten years follow-up of health and disability in people with acute traumatic hand injury: pain and cold sensitivity are long-standing problems. J Hand Surg Eur Vol. 2011 Sep;36(7):590-8. doi: 10.1177/1753193411408186. Epub 2011 May 18. PMID 21593072
- [Background] Craigen M, Kleinert JM, Crain GM, McCabe SJ. Patient and injury characteristics in the development of cold sensitivity of the hand: a prospective cohort study. J Hand Surg Am. 1999 Jan;24(1):8-15. doi: 10.1053/jhsu.1999.jhsu24a0008. PMID 10048510
- [Background] Novak CB, McCabe SJ. Prevalence of cold sensitivity in patients with hand pathology. Hand (N Y). 2015 Jun;10(2):173-6. doi: 10.1007/s11552-014-9694-y. PMID 26034426
- [Background] McCabe SJ, Mizgala C, Glickman L. The measurement of cold sensitivity of the hand. J Hand Surg Am. 1991 Nov;16(6):1037-40. doi: 10.1016/s0363-5023(10)80065-6. PMID 1748748
- [Background] Carlsson I, Cederlund R, Hoglund P, Lundborg G, Rosen B. Hand injuries and cold sensitivity: reliability and validity of cold sensitivity questionnaires. Disabil Rehabil. 2008;30(25):1920-8. doi: 10.1080/09638280701679705. PMID 19061118
- [Background] Ruijs AC, Jaquet JB, Daanen HA, Hovius SE. Cold intolerance of the hand measured by the CISS questionnaire in a normative study population. J Hand Surg Br. 2006 Oct;31(5):533-6. doi: 10.1016/j.jhsb.2006.04.013. Epub 2006 Jun 30. PMID 16808991
- [Background] Magistroni E, Ferriero G, Peri E, Parodi G, Massazza G, Franchignoni F. Psychometric properties of the Italian version of the Cold Intolerance Symptom Severity questionnaire in upper-extremity nerve repair. Eur J Phys Rehabil Med. 2019 Oct;55(5):627-633. doi: 10.23736/S1973-9087.19.05555-2. Epub 2019 Jan 8. PMID 30621369
- [Background] Tore NG, Gomussoy M, Oskay D. Validity and reliability of the Turkish version of the Cold Intolerance Symptom Severity Questionnaire. Turk J Med Sci. 2019 Aug 8;49(4):1221-1227. doi: 10.3906/sag-1808-170. PMID 30866612
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Background] Prinsen CAC, Mokkink LB, Bouter LM, Alonso J, Patrick DL, de Vet HCW, Terwee CB. COSMIN guideline for systematic reviews of patient-reported outcome measures. Qual Life Res. 2018 May;27(5):1147-1157. doi: 10.1007/s11136-018-1798-3. Epub 2018 Feb 12. PMID 29435801
- [Background] Polit DF, Beck CT. The content validity index: are you sure you know what's being reported? Critique and recommendations. Res Nurs Health. 2006 Oct;29(5):489-97. doi: 10.1002/nur.20147. PMID 16977646
- [Result] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735